CLINICAL TRIAL: NCT06739954
Title: Effectiveness of Dry Needling With or Without Mulligan Two Leg Rotation Technique on Pain, Range of Motion and Joint Dysfunction in Knee Osteoarthritis
Brief Title: Effectiveness of DN With or Without Mulligan Two Leg Rotation Technique on Pain ROM and Joint Dysfunction in KO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/773
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Combination Product: Mulligan's Two Leg Rotation technique
- Interventional group II (Active Comparator)
  Interventions: Diagnostic Test: Dry Needling

INTERVENTIONS:
Combination Product: Mulligan's Two Leg Rotation technique — The participants will undergo Mulligan's Two Leg Rotation technique, performing 10 repetitions with a 30-second hold for each repeat. There will be a 1-minute rest period between each stretch. The therapist positions themselves on the affected side of the supine patient lying on the treatment table and holds onto the side of the table with their hand on the opposite side. Both legs will be bent so that the feet are raised from the plinth. Maintaining the subject's shoulders on the bed, he gradually moves the subject's legs to the side, considering the restricted flexibility of the hamstring muscles. Once the patient reaches their maximum, the therapist applies extra pressure to sustain the posture for 30 seconds. Then, the legs are lowered to the plinth. A 1-minute interval was provided between each stretch, and the stretches were performed for a total of 10 repetitions. The identical technique is performed on the opposite side to address insufficient flexibility in the hamstrings.
  Arms: Interventional group I
Diagnostic Test: Dry Needling — The DN technique, based on previous research, involved slowly inserting and removing the needle in the muscle or tendon to elicit a specific response. This response could be a local twitch, a dull ache, a feeling of heaviness or distension, or the reproduction of the participant's symptoms. The needle is manipulated in and out of the targeted tissue five times every five minutes for a total of fifteen minutes. After the treatment, sterile gauze is applied and pressed on the DN site, and sterile non-stick pads are used to cover the treated areas. The number of needles used varied depending on the participant's condition. The knee muscles that will be included in the dry needling intervention are the Quadriceps and Hamstrings .
  Arms: Interventional group II

SUMMARY:
The objective of study is to determine the effectiveness of dry needling with or without mulligan two leg rotation technique on pain, range of motion and joint dysfunction in knee osteoarthritis. The study will be a single blinded randomized controlled trial conducted at the Physical Therapy Department of Hussain Memorial Hospital, focusing on the treatment of knee osteoarthritis in adults aged 40 to 80 years.

DETAILED DESCRIPTION:
The selection criteria will include patients with a confirmed diagnosis of knee osteoarthritis according to the Kellgren and Lawrence classification system, persistent symptoms for at least 6 months, and willingness to participate in the study. Exclusion criteria will include patients with other joint pathologies, severe psychiatric disorders, unstable medical conditions, or currently enrolled in another clinical trial. The sample size will be 40 patients, and divided into two groups, with Group A receiving dry needling combined with Mulligan two-leg rotation technique and Group B receiving only dry needling.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age 18-65 diagnosed with chronic coccydynia for at least 3 months were recruited.
* Participants who will be willing & able to adhere to the study protocol.
* Including participants who will be attending follow-up appointments & completing outcome measures.
* Participants who will be able to understand & provide written informed consent.
* Participants with a complete screening of other medical conditions and previous medical records.

Exclusion Criteria:

* Participants with previous surgery on the coccyx or lumbosacral spine, pregnancy or breastfeeding, history of bleeding disorders or anticoagulant use, active infection, or significant medical condition that could pose a safety risk during the procedures (GIB or CESI) was omitted.
* Patients above the age of 65 were eliminated to reduce confounding by age-related health concerns and to provide a more homogenous study population for more accurate treatment outcomes.
* Participants with neurological conditions affecting pain perception or sensation were excluded.
* Participants with known allergies to medications used in the study (local anesthetic, steroid for injections) were not part of the study.
* Participation in another interventional clinical trial within the past 3 months was not included.
* Participants who were unable to safely undergo fluoroscopy were also excluded.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  It is a tool used to measure pain intensity. It consists of a 10cm line with two endpoints representing 0, indicating 'no pain,' and 10, indicating 'pain as bad as it could possibly be.' Patients are asked to rate their current level of pain by marking the line accordingly. The distance in centimeters from the 'no pain marker' or zero to the marked point is measured using a ruler. This measurement provides a pain intensity score on a scale of 0 to 10. For example, a score of 6 out of 10 (or 6/10) indicates a pain level of 6.
Western Ontario and McMaster universities osteoarthritis (WOMAC) index | 12 Months
  This self-administered questionnaire was presented using a five-point ordinal scale with five categorical responses (numerical value of 0-4). WOMAC was designed to measure perceived pain, stiffness and dysfunction. High WOMAC scores reflect greater severity across the three measured domains. WOMAC has moderate-to-excellent reliability and validity to test pain, stiffness and function, especially in patients with hip or knee OA

CONTACTS AND LOCATIONS:
Locations (1):
- Ghurki trust and teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No